CLINICAL TRIAL: NCT06512818
Title: Effect of Psiguavin, a Bioactive Compound Derived From Psidium Guava, as Therapeutic Agent for Obesity Treatment
Brief Title: Effect of Psiguavin for Obesity Treatment (PSIGUAVIN)
Acronym: PSIGUAVIN
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Juan Jose Hernández Morante, Research Coordinator of the Faculty of Nursing Studies, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIO_HPC-2
Record Dates: First submitted 2023-09-20; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Obesity; Overweight or Obesity
Keywords: obesity; weight loss; pancreatic lipase; psiguavin
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Intervention Model Description: There wiil be two arms. One group will undergo the intervention with the bioactive compound psiguavin, and the other will follow a placebo-based treatment. Both groups will start and finish the project at the same time.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERVENTION WITH PSIDIUM GUAVA EXTRACT (Experimental): The volunteers in this group will undergo an intervention with a dose of 300 mg of psiguavin derived from Psidium guava extracts, three times a day, with each main meal.
  Interventions: Dietary Supplement: Psiguavin
- PLACEBO CONTROLLED INTERVENTION (Placebo Comparator): The volunteers in this group will undergo a placebo (microcellulose) with similar aspect than intervention, three times a day, with each main meal.
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Psiguavin — A purified guava extract will be used, enriched in psiguavin
  Other Names: Guava extract
  Arms: INTERVENTION WITH PSIDIUM GUAVA EXTRACT
Drug: Placebo — Capsules with the same characteristics that Psiguavin intervention but filled with a placebo compound
  Other Names: Placebo controlled intervention
  Arms: PLACEBO CONTROLLED INTERVENTION

SUMMARY:
The main objective of the project focuses on the study of the effectiveness of a functional component extracted from Psidium guava, psiguavin, as a potential inhibitor of pancreatic lipase and, therefore, as an adjuvant for the treatment of obesity.

That is, the aim is to verify from various experimental perspectives the effect of psiguavin on the activity of the enzyme pancreatic lipase (EC 3.1.1.3), which is the main enzyme responsible for the digestion of lipids from the diet. Our preliminary studies have shown that there is a strong interaction between psiguavin and the active center of pancreatic lipase; however, it is necessary to confirm these initial hypotheses through a clinical trial. Taking into account that the usefulness of this compound is based on the reduction of dietary calorie intake, in order to confirm its therapeutic usefulness, a clinical trial will be proposed.

To this end, the following specific objective is defined, which is intended to be achieved with the execution of the project:

• Evaluate the effect of psiguavin on weight loss of people with overweight/obese people.

DETAILED DESCRIPTION:
The latest data published by the World Health Organization (WHO) report that overweight and obesity are the most prevalent diseases worldwide. In 2016, 39% of adults worldwide were overweight, and 13% were obese. Although there are many factors involved in the development of obesity, an excessive intake of calories, especially in the form of fat, and a sedentary lifestyle are still considered the key factors for the development of overweight.

Currently, the standard treatment or therapy for obesity is the modification of habits or lifestyles, reducing energy intake through low-calorie diets, and increasing energy expenditure with physical activity programs. The problem is that the effectiveness of these interventions is usually very modest, especially in the long term. On certain occasions (such as when weight losses are very small), in addition to this therapy that we can define as "conventional", certain drugs can be prescribed to reduce caloric intake and improve the effectiveness of the dietary intervention.

There are various drugs approved by the EMA and the AEMPS for the treatment of obesity: on the one hand, there are centrally acting agents such as the naltrexone-bupropion combination. On the other hand, peripherally acting agents, such as liraglutide or orlistat, have shown greater effectiveness for weight loss. Orlistat (Xenical®) is the best-selling obesity drug in the world, and is the only drug approved for adolescents; Its effectiveness is similar to other drugs, but it is safer because its adverse effects are related to gastrointestinal alterations, such as fecal urgency, fecal incontinence, flatus, steatorrhea, among others, which are frequently the cause of abandonment of this drug. treatment. For all these reasons, it seems evident that the most appropriate treatment for addressing obesity would be through a mechanism similar to that of orlistat, and if possible with greater effectiveness and fewer adverse effects.

Our previous in silico and in vitro studies have shown that the bioactive component of guava, psiguavin, has pharmacological characteristics very similar to orlistat, which is why we considered this clinical trial to confirm, in vivo, these previous data.

Psiguavin is a compound from the family of hydrolyzable tannins extracted from guava (Psidium guajava). This compound has been used in traditional botany for the treatment of disorders related to the accumulation of liver fat induced by excess sugars. Despite this, there are no clear bibliographic references on the compound's potential for use as a bioactive compound for application in the treatment of obesity.

To this end, a double-arm, double-blind, randomized, placebo-controlled study will be carried out to analyze weight loss in overweight/obese patients during a period of 3 months of treatment plus one year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 65 years old
* Having a BMI between 25 and 40
* Voluntarily taking part in the study

Exclusion Criteria:

* Have been on a diet for at least 6 months before the start of the study.
* Taking chronic medication that can alter metabolism (thyroid drugs, corticosteroids, etc.)
* Having a contraindication for guava
* Having an intestinal chronic disease
* Being pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-08 (Estimated); Primary Completion 2026-12-19 (Estimated); Study Completion 2027-12-19 (Estimated)

PRIMARY OUTCOMES:
Percentage of body weight loss | At three months from baseline and after one-year of follow-up
  It will be calculated by subtracting the initial weight less to the final weight, divided by the initial weight and multiplied by 100.
Percentage of body fat loss | At three months from baseline and after one-year of follow-up
  Meaured by impedance, the change in final fat percentage with respect to the initial value will be calculated.

SECONDARY OUTCOMES:
Metabolic syndrome status | At three months from baseline and after one-year of follow-up
  The diagnosis of metabolic syndrome will be analyzed according to the IDF criteria.
Plasma total cholesterol levels | At three months from baseline and after one-year of follow-up
  Changes in total cholesterol levels will analyzed determining the plasma cholesterol at the end of the intervention minus baseline cholesterol (measured in mg/dl)
Plasma triglyceride levels | At three months from baseline and after one-year of follow-up
  Changes in triglyceride levels will analyzed determining the plasma triglycerides at the end of the intervention minus baseline triglycerides (measured in mg/dl)
Fasting plasma glucose levels | At three months from baseline and after one-year of follow-up
  Changes in fasting glucose levels will analyzed determining the plasma fasting glucose at the end of the intervention minus baseline fasting plasna (measured in mg/dl)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing. Catholic University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided